CLINICAL TRIAL: NCT06033092
Title: Low Dose TamOxifen and LifestylE Changes for bReast cANcer prevenTion: a Randomized Phase II Biomarker Trial in Subjects at Increased Risk
Brief Title: Low Dose TamOxifen and LifestylE Changes for bReast cANcer prevenTion
Acronym: TOLERANT
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: European Institute of Oncology (Other)
Collaborators: Ente Ospedaliero Ospedali Galliera (Other); Istituto Oncologico Veneto IRCCS (Other); Istituto Nazionale Tumori IRCCS - Fondazione G. Pascale (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: UID 3751; 2023-503994-39-00 (Other: EU CT number)
Record Dates: First submitted 2023-08-23; First posted 2023-09-13 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: BRCA Mutation; PALB2 Gene Mutation; Ductal Carcinoma in Situ; Lobular Carcinoma in Situ; ATM Gene Mutation; CHEK2 Gene Mutation; CDH1 Gene Mutation; RAD51C Gene Mutation; RAD51D Gene Mutation
Keywords: Low Dose Tamoxifen; Intermittent Caloric Restriction; Sex Hormone Binding Globulin; Lifestyle
MeSH Terms: conditions — Carcinoma, Intraductal, Noninfiltrating; Breast Carcinoma In Situ | interventions — Tamoxifen; Tablets

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Low dose tamoxifen (Active Comparator): Tamoxifen 10 mg (1 tablet) every other day for 6 months.
  Interventions: Drug: Tamoxifen 10 mg Tablet
- Low dose tamoxifen + Intermittent Caloric Restriction (Active Comparator): Tamoxifen 10 mg (1 tablet) every other day for 6 months + 5:2 diet (5 days/week at regular energy intake+2 days a week at an average 75% energy deficit)
  Interventions: Drug: Tamoxifen 10 mg Tablet; Other: Intermittent caloric restriction
- Lifestyle intervention (Placebo Comparator): Step counter device
  Interventions: Behavioral: Step counter Device
- Lifestyle Intervention + Intermittent Caloric Restriction (Active Comparator): Step counter device + 5:2 diet (5 days/week at regular energy intake+2 days a week at an average 75% energy deficit)
  Interventions: Other: Intermittent caloric restriction; Behavioral: Step counter Device

INTERVENTIONS:
Drug: Tamoxifen 10 mg Tablet — One tablet of Tamoxifen 10 mg every other day for 6 months
  Other Names: Low dose tamoxifen
  Arms: Low dose tamoxifen; Low dose tamoxifen + Intermittent Caloric Restriction
Other: Intermittent caloric restriction — "5:2 diet": 5 days a week at regular energy intake and 2 days/week at 75% energy deficit (diet will be restricted at 500-800 kcal corresponding to a 75% reduction compared to normal size)
  Arms: Lifestyle Intervention + Intermittent Caloric Restriction; Low dose tamoxifen + Intermittent Caloric Restriction
Behavioral: Step counter Device — Participants will receive personal advice on healthy lifestyle and a step counter
  Arms: Lifestyle Intervention + Intermittent Caloric Restriction; Lifestyle intervention

SUMMARY:
Circulating levels of Sex Hormone Binding Globulin (SHBG) are significantly associated with a decreased risk of breast cancer.

The main aim of this clinical trial is to verify whether Low Dose Tamoxifen (LDT) increases circulating levels of SHBG more than lifestyle intervention (LI) with or without intermittent caloric restriction (ICR) after 6 months in women at increased risk of breast cancer (i.e., healthy participants carriers of a germline pathogenic/likely pathogenetic variant in at least one of the following genes: BRCA1, BRCA2, PALB2, ATM, CHEK2, CDH1, RAD51C or RAD51D, or with > 5% breast cancer risk at 10 years, using the Tyrer Cuzick or the Breast Cancer Surveillance Consortium Risk models or with a recently resected intraepithelial neoplasia of the breast (IEN).

The secondary aims are:

* to verify whether ICR significantly modulates primary and secondary endpoints such as Homeostasis Model Assessment (HOMA) index, immune and inflammatory markers, lipid profile, Adiponectin/Leptin (A/L) ratio, quality of life (QoL), Body mass index (BMI), fat body composition, safety and toxicity;
* to verify whether LDT significantly modulates secondary endpoints, such as HOMA-index, immune and inflammatory markers, lipid profile, A/L ratio, QoL, BMI, fat body composition, safety and toxicity;
* to investigate differences in microbiome composition by arms and the effect of changes in microbiome on QoL taking into account circulating biomarkers, cytokines, immune modulators, and inflammatory proteins in serum;
* to investigate MD (Mammographic Breast Density) changes by LDT vs. LI, with or without ICR. This aim will be performed in a subgroup of participants (not all the participants will undergo mammography due to younger age).

DETAILED DESCRIPTION:
Italian, multicenter, phase II, biomarker trial. A total of 200 women aged 18-70 years will be randomly assigned (1:1:1:1) to one of the four intervention arms Arm 1: Low dose Tamoxifen (LDT) i.e. 10 mg every other day; Arm 2: Low dose Tamoxifen (LDT) + Intermittent Caloric Restriction (ICR); Arm 3: Lifestyle intervention (LI) using a step counter; Arm 4: Lifestyle intervention (LI) using a step counter + Intermittent Caloric Restriction (ICR).

Participants will be stratified by center and by disease status (high risk vs. previous IEN) and intervention will last six months for all arms.

ELIGIBILITY:
Inclusion Criteria:

1. Women between 18 and 70 years old;
2. Healthy participants carriers of a germline pathogenic/likely pathogenetic variant in at least one of the following genes BRCA1, BRCA2, PALB2, ATM, CHEK2, CDH1, RAD51C or RAD51D, or

   > 5% breast cancer risk at 10 years, using the Tyrer Cuzick or the Breast Cancer Surveillance Consortium Risk models, or

   with previous diagnosis of intraepithelial neoplasia (surgery for ADH, LCIS, ER positive DCIS) within the last 3 years;
3. Ability to understand and the willingness to sign a written informed consent document;
4. Eastern Cooperative Oncology Group (ECOG) Performance Status ≤1;

5a. For high-risk strata: A negative mammogram or any radiological image based on age and center protocol screening within 6 months before baseline visit;

5b. For IEN Strata: A negative mammogram within 12 months before baseline visit;

6. A negative transvaginal ultrasound within 6 months before baseline visit.

Exclusion Criteria:

1. Diagnosis of ER-negative (<10%) DCIS, or history of invasive breast cancer;
2. Previous treatment with SERMs or any other hormonal treatment for breast neoplasms;
3. BMI < 18.5 Kg/m2 and/or Malnutrition Universal Screening Tool (MUST) score ≥2 and/or any current or past eating disorders;
4. Any diagnosis of invasive neoplasia, except non-melanoma skin cancer, in the previous 5 years;
5. Any tamoxifen contraindications (abnormal liver function, previous ischemic heart disease, endometrial disorder, previous deep venous thrombosis, history of pulmonary embolus, current or suspected glaucoma, retinopathy and cataract);
6. Current use of warfarin or other anticoagulant drugs
7. Bilateral mastectomy;
8. Pregnancy or desire to become pregnant in the subsequent 9 months after treatment cessation;
9. Diabetes or any other clinical condition that at the investigator's discretion contraindicates the proposed intervention.
10. No hormonal contraception is allowed during study intervention. Non-hormonal methods will be advised for women of childbearing potential (WOCBP)

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 200 (Estimated)
Dates: Start 2024-06-21 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Post intervention levels of circulating binding globulin | Through study completion, an average of 6 months
  Sex hormone binding globulin level after 6 months of intervention

CONTACTS AND LOCATIONS:
Overall Officials: Bernardo Bonanni, MD, Principal Investigator — Istituto Europeo di Oncologia
Locations (4):
- Italy (4):
  - E.O. Galliera, Genoa
  - Istituto Europeo di Oncologia, Milan
  - Istituto Nazionale Tumori G. Pascale, Napoli
  - Istituto Oncologico Veneto, Padua

REFERENCES:
- [Derived] Guerrieri-Gonzaga A, Serrano D, Gnagnarella P, Johansson H, Zovato S, Nardi M, Pensabene M, Buccolo S, DeCensi A, Briata IM, Pistelli L, Sansone C, Mannucci S, Aristarco V, Macis D, Lazzeroni M, Aurilio G, Accornero CA, Gandini S, Bonanni B. Low dose TamOxifen and LifestylE changes for bReast cANcer prevention (TOLERANT study): Study protocol of a randomized phase II biomarker trial in women at increased risk for breast cancer. PLoS One. 2024 Sep 3;19(9):e0309511. doi: 10.1371/journal.pone.0309511. eCollection 2024. PMID 39226292